CLINICAL TRIAL: NCT03212534
Title: A Randomized Clinical Trial of a Mortality Prediction Algorithm
Brief Title: Inpatient Mortality Prediction Algorithm Clinical Trial (IMPACT)
Acronym: IMPACT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This trial did not start. No participants enrolled
Sponsor: Dascena (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-22319
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Decompensation, Heart; Decompensation; Heart, Congestive; Death
Keywords: Dascena; patient mortality; machine learning; algorithm; diagnostic
MeSH Terms: conditions — Heart Failure; Death; Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prediction Algorithm (Experimental)
  Interventions: Other: Patient mortality prediction
- Control (No Intervention)

INTERVENTIONS:
Other: Patient mortality prediction — Healthcare provider is notified of patient mortality prediction.
  Arms: Prediction Algorithm

SUMMARY:
Through the mapping of retrospective patient data into a discrete multidimensional space, a novel algorithm for homeostatic analysis, was built to make outcome predictions. In this prospective study, the ability of the algorithm to predict patient mortality and influence clinical outcomes, will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the participating units will be eligible.

Exclusion Criteria:

* All patients younger than 18 years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | Through study completion, an average of 30 days

SECONDARY OUTCOMES:
Hospital length of stay | Through study completion, an average of 30 days

OTHER OUTCOMES:
Hospital readmission | Through study completion, an average of 30 days
ICU length of stay | Through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: David Shimabukuro, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Moffit-Long Hospital, San Francisco, California, United States

REFERENCES:
- [Background] Desautels T, Calvert J, Hoffman J, Mao Q, Jay M, Fletcher G, Barton C, Chettipally U, Kerem Y, Das R. Using Transfer Learning for Improved Mortality Prediction in a Data-Scarce Hospital Setting. Biomed Inform Insights. 2017 Jun 12;9:1178222617712994. doi: 10.1177/1178222617712994. eCollection 2017. PMID 28638239
- [Background] Calvert J, Mao Q, Rogers AJ, Barton C, Jay M, Desautels T, Mohamadlou H, Jan J, Das R. A computational approach to mortality prediction of alcohol use disorder inpatients. Comput Biol Med. 2016 Aug 1;75:74-9. doi: 10.1016/j.compbiomed.2016.05.015. Epub 2016 May 24. PMID 27253619
- [Background] Calvert JS, Price DA, Barton CW, Chettipally UK, Das R. Discharge recommendation based on a novel technique of homeostatic analysis. J Am Med Inform Assoc. 2017 Jan;24(1):24-29. doi: 10.1093/jamia/ocw014. Epub 2016 Mar 28. PMID 27026611
- [Background] Calvert J, Mao Q, Hoffman JL, Jay M, Desautels T, Mohamadlou H, Chettipally U, Das R. Using electronic health record collected clinical variables to predict medical intensive care unit mortality. Ann Med Surg (Lond). 2016 Sep 6;11:52-57. doi: 10.1016/j.amsu.2016.09.002. eCollection 2016 Nov. PMID 27699003